CLINICAL TRIAL: NCT00524862
Title: Selective Strategy to Manage Arrhythmia Risk and Therapy With ICD
Brief Title: Standard Drug Therapy vs. Implanted Defibrillator for Primary Prevention of Sudden Cardiac Death
Acronym: SMART-ICD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Unity Health Toronto (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06368
Record Dates: First submitted 2007-08-29; First posted 2007-09-05 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Heart Disease; Congestive Heart Failure; Ventricular Dysfunction; Low Cardiac Output; Sudden Cardiac Death
Keywords: Implantable Cardioverter Defibrillator; Ejection Fraction; QRS duration
MeSH Terms: conditions — Coronary Disease; Heart Failure; Ventricular Dysfunction; Cardiac Output, Low; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other)
  Interventions: Drug: Optimized medical therapy
- 2 (Other)
  Interventions: Device: Implantable Cardioverter Defibrillator

INTERVENTIONS:
Drug: Optimized medical therapy — Beta Blockers, ACE inhibitor or ARB, loop diuretics and/or spironolactone as appropriate, statin if indicated, aspirin and/or warfarin if indicated
  Arms: 1
Device: Implantable Cardioverter Defibrillator — an implanted device, called a defibrillator, which monitors heart rhythm and treats life-threatening rhythms accordingly
  Other Names: ICD
  Arms: 2

SUMMARY:
Recent ACC/AHA/ESC guidelines recommend prophylactic ICD implantation in most patients with coronary heart disease and LVEF < 40%. Current Canadian guidelines recommend ICDs for primary prophylaxis in CAD patients with LVEF < 30% (Class I recommendation). There are very sparse data to recommend ICD implantation in patients with EF between 30 and 40 %. This study will randomize patients with CHD and an EF between 30 and 40% to ICD therapy vs. No ICD therapy. The primary outcome is mortality and the study is powered as a non-inferiority trial to test the hypothesis that mortality in patients with no ICD is not more than 1% greater (absolute yearly increase) than patients receiving an ICD.

ELIGIBILITY:
Inclusion Criteria:

* documented chronic coronary heart disease (prior MI and/or angiographically documented CAD), > 40 days post the most recent MI;
* LVEF < 40% (by MUGA) and NYHA functional class II or III at time of assessment OR LVEF ≤ 35 % (by MUGA) and NYHA functional class I, II or III at time of assessment
* Judged to have a reasonable expectation of survival with a good functional status for more than 1 year, as well as receiving optimum, guideline recommended therapy for coronary artery disease and heart failure (or demonstrated intolerance or contraindications to such therapy).
* Age ≥ 18 years; no upper age limitation.

Exclusion Criteria:

* Prior cardiac arrest, sustained VT or VF, or unexplained syncope.
* Attempted VT / VF induction at electrophysiological study.
* Need for a cardiac resynchronization therapy (CRT) device.
* Enrollment in another interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | minimum 1 year follow-up (maximum 6 year)

SECONDARY OUTCOMES:
1. Presumed arrhythmic (sudden death) mortality. 2. Major morbidity which includes mortality, hospitalization and major device complications | minimum 1 year; maximum 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dorian, MD, Study Chair — Unity Health Toronto; Andreas Laupacis, MD, Study Director — Li Ka Shing Knowledge Institute at St. Michael's Hospital; Douglas Lee, MD, Study Director — Institute for Clinical Evaluatuve Sciences; Kevin Thorpe, MSc, Study Director — Li Ka Shing Knowledge Institute at St. Michael's Hospital; Marta Gadacz, MSc, Study Director — Unity Health Toronto
Locations (10):
- Canada (10):
  - Hamilton Health Sciences - Hamilton General, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences - University Campus, London, Ontario
  - Trillium Health Centre - Mississauga, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Rouge Valley Health System - Centenary, Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario